CLINICAL TRIAL: NCT03807375
Title: Evaluation of the Effect of CPAP and Mask Ventilation on Preoxygenation Time in Bariatric Surgery
Brief Title: The Comparison of the Methods Applied in Bariatric Surgery in Terms of Preoxygenation Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ilkay baran akkuş, principle investigator, Ankara Diskapi Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: preoxygenation
Record Dates: First submitted 2019-01-10; First posted 2019-01-16 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-01

CONDITIONS: Time to Reach 90% Endtidal Oxygen During Preoxygenation
Keywords: CPAP(Continuous Positive Airway Pressure); Standard preoxygenation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP (Other): During preoxygenation, the ventilator device will be placed in spontaneous mode and set as CPAP: 5 cmH2O. The process will continue until the end-tidal O2 concentration ≥ 90% is removed.
  Interventions: Other: CPAP preoxygenation
- standard preoxygenation (No Intervention): During the preoxygenation, the ventilator device will be put in spontaneous mode and the procedure will continue until the End-tidal O2 concentration ≥90% is removed without additional pressure.

INTERVENTIONS:
Other: CPAP preoxygenation — During preoxygenation, the ventilator device will be placed in spontaneous mode and set as CPAP: 5 cmH2O.
  Arms: CPAP

SUMMARY:
The aim of the study was to evaluate the preoxygenation time by observing patients undergoing preoxygenation with CPAP (Continuous Positive Airway Pressure) and Mask Ventilation in the clinic.

DETAILED DESCRIPTION:
Criteria for inclusion in the study:

Planned elective bariatric surgery under general anesthesia ASA 1-2 class Between 20-50 years 50 patients

1. Group: Patients undergoing CPAP (Continuous Positive Airway Pressure) during preoxygenation will be included.
2. Group: Patients undergoing preoxygenation without CPAP will be included

In both groups, the time from the anesthesia device to the endtidal O2 90% and the endtidal CO2 value in this order will be recorded.

Heart rate, blood pressure, endtidal O2 and CO2 values will be recorded during preoxygenation and after intubation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Patients between the ages of 20 and 50 years
  2. American Society of Anesthesiologists I, II or III
  3. Patients with body mass index of 40 and over

Exclusion Criteria:

1. cardiopulmonary disease
2. patients with previous abdominal or thoracic surgery or cerebrovascular disease
3. story of intracranial hypertension or epilepsy
4. patients with a story of difficult tracheal intubation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Prevention of desaturation during intubation | 5 minutes
  Prevent desaturation of the apnea period during endotracheal intubation in bariatric surgery
prevention of side effects of hypoxia | 10 minutes
  hypoxia-induced arrhythmia hypotension tachycardia

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Yildirim Beyazit Training Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouroche G, Bourgain JL. Preoxygenation and general anesthesia: a review. Minerva Anestesiol. 2015 Aug;81(8):910-20. Epub 2015 Jun 5. PMID 26044934
- [Result] Nimmagadda U, Salem MR, Crystal GJ. Preoxygenation: Physiologic Basis, Benefits, and Potential Risks. Anesth Analg. 2017 Feb;124(2):507-517. doi: 10.1213/ANE.0000000000001589. PMID 28099321